CLINICAL TRIAL: NCT04723550
Title: Impact of Telemedicine on Young and Middle-aged Obese Patients With Type 2 Diabetes Mellitus During COVID-19 Pandemic
Brief Title: COVID-19 Lockdown Related Telemedicine for Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wenwen Yin (Other)
Responsible Party: Sponsor-Investigator, Wenwen Yin, M.D., Xuzhou No.1 Peoples Hospital
Organization: Xuzhou No.1 Peoples Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NO.2020QN80
Record Dates: First submitted 2021-01-21; First posted 2021-01-25 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; COVID-19 lockdown; Telemedicine; Obesity; Young and middle-aged
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine (Experimental): Diabetes education and support by telemedicine
  Interventions: Device: Hospital telemedicine management system
- Usual care (Active Comparator): Diabetes education and support in person
  Interventions: Other: Usual care

INTERVENTIONS:
Device: Hospital telemedicine management system — Patients upload data of blood glucose, diet and exercise. Then doctors guide patients' diet, exercise and medication adjustment through the telemedicine system.
  Arms: Telemedicine
Other: Usual care — Outpatient/telephone follow-up：continued care, as usual, from their primary care provider through out duration of action 6 months intervention period
  Arms: Usual care

SUMMARY:
At present, in order to cope with the global pandemic of the COVID-19 virus, governments have introduced corresponding measures, COVID-19 lockdown is one of the most important measures. However, lockdown makes the management of chronic diseases (such as type 2 diabetes) more difficult, and telemedicine may be one of the solutions. We hope to explore the effect of telemedicine on blood glucose control and other prognostic indicators of young and middle-aged obese patients with type 2 diabetes who will experience isolation control.

DETAILED DESCRIPTION:
We recruit patients with type 2 diabetes who need to be isolated due to the COVID-19 epidemic, Our study will include young and middle-aged obese patients. The lockdown period is 21 days. The patients will be randomly divided into two groups with a total follow-up time of 6 months. One group is the telemedicine intervention group, and the other group is the routine follow-up control group. The intervention group used the hospital telemedicine management system to upload blood glucose values (fasting and 2h after three meals), food intake of three meals, and exercise volume (Data collection frequency: first three months, 4 times/week; 4-6 Month, 2 times/week).Doctors will collect data from hospital telemedicine management system to guide patients on diets, exercise, and medication adjustments. The control group will be followed up by telephone/outpatient clinic every 1 week. (only telephone follow-up will be conducted during the lockdown period) Then doctors will collect their blood glucose values.(fasting and 2h after three meals) Based on the data collected, The doctors will provide lifestyle guidance to the patients on the telephone or face to face. The clinical data of the two groups of patients will be collected at baseline, 22 days, 3 months, and 6 months respectively. (HbA1c, fasting blood glucose(FBG), blood glucose 2 hours after breakfast, blood pressure, Body Mass Index(BMI), waist-to-hip ratio, total cholesterol(TC), triglyceride(TG), high-density lipoprotein cholesterol(HDL-C), low-density lipoprotein cholesterol(LDL-C), Blood Urea Nitrogen(BUN), serum creatinine(Scr), e-GFR, Self-rating Depression Scale, frequency of hypoglycemia，and Cost effectiveness) The clinical data will be statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of Type 2 diabetes for more than 6 months
* 7.0%<HbA1c<10.0%
* Quarantine for 21 days due to COVID-19 outbreak related reasons
* age: 18 ~ 55 yrs
* BMI≥24
* Be able use smart phones and the Internet

Exclusion Criteria:

* Insulin pump users
* For female subjects: pregnancy or lactation, or subject may become pregnant during the study
* Patient who underwent obesity surgery to the exclusion of a gastric band, loosened or removed for more than a year
* Patients diagnosed with COVID-19 infection
* Have severe complications (chronic heart disease, cerebrovascular disease, diagnosed HIV/AIDS, cancer, emphysema, chronic liver or kidney disease) that would affect the subjects' ability to follow the tailored advice

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-11-05 (Estimated); Study Completion 2022-01-05 (Estimated)

PRIMARY OUTCOMES:
Glucose control (HbA1c levels) | Baseline, 22days,3 months and 6 months
  Change in HbA1c among control and telemedicine groups from baseline to 6 months

SECONDARY OUTCOMES:
Change in FBG | Baseline, 22days,3 months and 6 months
  Change in FBG among control and telemedicine groups from baseline to 6 months
Change in Blood glucose 2 hours after breakfast | Baseline, 22days,3 months and 6 months
  Change in Blood glucose 2 hours after breakfast among control and telemedicine groups from baseline to 6 months
Change in Blood pressure | Baseline, 22days,3 months and 6 months
  Change in Blood pressure among control and telemedicine groups from baseline to 6 months
Body mass BMI changes | Baseline, 22days,3 months and 6 months
  Comparison of BMI changes among control and telemedicine groups from baseline to 6 months
Change in waist-to-hip ratio | 6 months
  Comparison of waist-to-hip ratio changes among control and telemedicine groups from baseline to 6 months
Change in biological parameter: TC | Baseline, 22days,3 months and 6 months
  Variation between baseline to 6 months of Biological parameter among control and telemedicine groups: TC
Change in biological parameter: TG | Baseline, 22days,3 months and 6 months
  Variation between baseline to 6 months of Biological parameter among control and telemedicine groups: TG
Change in biological parameter: HDL-C | Baseline, 22days,3 months and 6 months
  Variation between baseline to 6 months of Biological parameter among control and telemedicine groups: HDL-C
Change in biological parameter: BUN | Baseline, 22days,3 months and 6 months
  Variation between baseline to 6 months of Biological parameter among control and telemedicine groups: BUN
Change in biological parameter: Scr | Baseline, 22days,3 months and 6 months
  Variation between baseline to 6 months of Biological parameter among control and telemedicine groups: Scr
Change in biological parameter: e-GFR | Baseline, 22days,3 months and 6 months
  Variation between baseline to 6 months of Biological parameter among control and telemedicine groups: e-GFR

OTHER OUTCOMES:
Change in scores measured by Self-rating Depression Scale | Baseline, 22days,3 months and 6 months
  Self-rating Depression Scale includes 20 items in four dimensions of psychological disorders, namely, psychotic emotional symptoms, somatic disorders, psychomotor disorders, and depression. The maximum value of SDS is 50 points. A lower total score means a better situation in terms of depression and vice versa
Number of hypoglycemia events | 6 months
  Hypoglycemia events for telemedicine group versus control group
Cost effectiveness | 6 months
  The objectives are to compare the results of the study in terms of cost and cost-effectiveness of these two strategies

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology, Xuzhou NO.1 Peoples Hospital, Xuzhou, Jiangsu, China

REFERENCES:
- [Derived] Yin W, Liu Y, Hu H, Sun J, Liu Y, Wang Z. Telemedicine management of type 2 diabetes mellitus in obese and overweight young and middle-aged patients during COVID-19 outbreak: A single-center, prospective, randomized control study. PLoS One. 2022 Sep 29;17(9):e0275251. doi: 10.1371/journal.pone.0275251. eCollection 2022. PMID 36174028